CLINICAL TRIAL: NCT00774254
Title: Participant Reactions to Disease Risk Information
Brief Title: Reactions to Disease Risk Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 090009; 09-HG-0009
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: Virtual Reality Technology; Communication; Doctor-Patient Communication
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: A; Behavioral: B

INTERVENTIONS:
Behavioral: A — Intervention
Behavioral: B — Intervention

SUMMARY:
This study is part of an effort to learn about interactions between doctors and patients. The study will use virtual reality technology to examine how patients and doctors interact when they discuss disease risks.

Men and women between the ages of 25 and 40 who have access to the Internet and were born and raised in the United States may be eligible for this study. Participants will be recruited from the Washington D.C. area.

Participants undergo the following procedures:

* Complete an online questionnaire about their health-related background, family health history, cancer risk perceptions, and demographic information (e.g., age, marital status, education, etc.).
* Participate in activities in a virtual reality environment in which they interact with a virtual doctor in a virtual clinical scenario. For this experiment, participants wear a head-mounted display that allows them to see the virtual world images.
* Fill out a second questionnaire after completing the virtual reality activities. This questionnaire includes information on the participants virtual reality experience, the information provided in the experience, and questions about themselves and their background.

DETAILED DESCRIPTION:
This study will investigate interactions between doctors and patients regarding risks of common, complex diseases using virtual reality technology.

Men and women between the ages of 25 and 40 who have access to the Internet and were born and raised in the United States may be eligible for this study. Participants will be recruited from the Washington D.C. area.

Study subjects complete two phases. The first phase is to complete an online questionnaire about their heath-related background, family health history, cancer risk perceptions, and demographic information using a secure survey website. The second phase involves interacting with a virtual doctor in a virtual environment clinical scenario, followed by completion of a second questionnaire. While in the virtual environment, participants wear a head-mounted video unit that allows them to see elements of the environment. The activities in the virtual environment take about 15 minutes. The total time for the study is about 60 minutes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Self-reported ability to speak, read, and write in English.
* Self identifying as African-American or Black
* Having been born and raised in the U.S.
* Not having been diagnosed with any of the diseases used in the experiment.
* Being between 25 and 40 years of age.
* Having access to the Internet.
* Both men and women will be included in the study.

EXCLUSION CRITERIA:

* Individuals below the age of 25 because they might not yet have completed their education and those above the age of 40 because they might have less familiarity with interactive technologies than younger individuals.
* Because the study will utilize virtual reality technology, individuals who are particularly susceptible to motion sickness will be excluded.
* All individuals with epilepsy, low vision, hearing problems, and vestibular disorders (e.g., vertigo) will be excluded from the study for safety reasons.
* We will re-screen for safety exclusion criteria when participants arrive to participate in the in-person portion of the study.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2009-06-16 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-09-30 (Actual)

PRIMARY OUTCOMES:
Risk Perception | ongoing
  The objective of the proposed study is to examine a cognitive bias known as anchoring and adjustment that may occur during provider-patient interactions, such as during provision of risk information for common, complex diseases that have both genetic and behavioralcomponents.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Loomis JM, Blascovich JJ, Beall AC. Immersive virtual environment technology as a basic research tool in psychology. Behav Res Methods Instrum Comput. 1999 Nov;31(4):557-64. doi: 10.3758/bf03200735. PMID 10633974
- [Background] Bailenson JN, Blascovich J, Beall AC, Loomis JM. Interpersonal distance in immersive virtual environments. Pers Soc Psychol Bull. 2003 Jul;29(7):819-33. doi: 10.1177/0146167203029007002. PMID 15018671
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-HG-0009.html